CLINICAL TRIAL: NCT02532595
Title: Trigger Point Dry Needling, Manual Therapy and Exercise vs Manual Therapy and Exercise For the Management of Achilles Tendinopathy
Brief Title: TDN, Manual Therapy and Exercise For the Management of Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03261504F
Record Dates: First submitted 2015-08-14; First posted 2015-08-26 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2020-01

CONDITIONS: Achilles Tendon Injury
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 manual therapy and exercise (Active Comparator): manual therapy with soft tissue mobilization to trigger points in the gastrocnemius, soleus, and tibialis posterior; exercise including stretching, concentric and eccentric exercises to the hip, triceps surae, tibialis posterior and foot intrinsics.
  Interventions: Procedure: manual therapy and exercise
- Group 2 TDN, manual therapy and exercise (Experimental): trigger point dry needling (TDN) to trigger points in the gastrocnemius, soleus and tibialis posterior; manual therapy with soft tissue mobilization to trigger points in the gastrocnemius, soleus, and tibialis posterior; exercise including stretching, concentric and eccentric exercises to the hip, triceps surae, tibialis posterior and foot intrinsics.
  Interventions: Procedure: manual therapy and exercise; Procedure: trigger point dry needling

INTERVENTIONS:
Procedure: manual therapy and exercise — soft tissue mobilization, stretches, concentric and eccentric strengthening
Procedure: trigger point dry needling — trigger point dry needling to trigger points located in the gastrocnemius, soleus and tibialis posterior
  Arms: Group 2 TDN, manual therapy and exercise

SUMMARY:
Conflicting evidence exists regarding the recommendations from the Orthopaedic section of the American Physical Therapy Association for treatment of Achilles tendinitis. Trigger point dry needling is effective in reducing pain in several body regions, but no published (TDN) studies are found reporting the effect on Achilles tendinopathy. The purpose of this study is to investigate whether a treatment program performed including TDN, manual therapy and exercise will result in a significant improvement in pain, strength and function compared to a treatment program including manual therapy and exercise for Achilles tendinopathy. Subjects with Achilles tendinopathy that receive treatment including TDN, manual therapy and exercise will demonstrate a significant improvement in pain, strength and functional outcomes compared to the group that receives manual therapy and exercise.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, pretest-posttest control group design comparing the effect of TDN, manual therapy and exercise to manual therapy and exercise on human subjects with Achilles tendinopathy following eight treatments in four weeks and a follow up examination at three months.

ELIGIBILITY:
Inclusion Criteria:

1. pain onset greater than 4 weeks
2. primary region of pain 2-6 cm proximal to the insertion on the calcaneus
3. read and write in english

Exclusion Criteria:

1. Fear of needles or unwilling to have needling performed due to fear or personal beliefs.
2. Vascular or sensory disturbances in the lower leg which include but is not limited to injury to the nerve root or peripheral nerve in the affected lower leg, inflammatory diseases, bleeding or clotting disorders, lymphedema, peripheral vascular or peripheral arterial disease. Diabetes is included in this group due to the progressive changes to the sensation and circulation in the lower extremities.
3. Recent infection.
4. Previous surgery to the foot/ankle.
5. Steroid by injection or transdermal delivery to the posterior heel within three months.
6. Full rupture of the Achilles tendon.
7. Pregnant or may be pregnant.
8. Participants with a work related injury insured by the bureau of worker's compensation or involved in litigation related to injury of the lower leg, foot or ankle.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Activity Level from baseline with the Functional Ankle Ability Measure | 4 weeks
Change in Functional Activity Level from baseline with the Functional Ankle Ability Measure | 3 months
Change in Pain from Baseline with the Numeric Pain Rating Scale | 4 weeks
Change in Pain from Baseline with the Numeric Pain Rating Scale | 3 months
Change in Fear of Activity from baseline with the Tampa Scale of Kinesiophobia | 4 weeks
Change in Fear of Activity from baseline with the Tampa Scale of Kinesiophobia | 3 months
Change in Pain from baseline with the Global Rating of Change | 4 weeks
Change in Pain from baseline with the Global Rating of Change | 3 months
Change in Pain from baseline with the Pain Pressure Threshold Measure | 4 weeks
  Primary site of pain on the Achilles tendon. All measurements taken with the Wagner FPK 20 Algometer.
Change in Pain from baseline with the Pain Pressure Threshold Measure | 3 months
  Primary site of pain on the Achilles tendon. All measurements taken with the Wagner FPK 20 Algometer.
Change in strength from baseline with the Muscle Endurance Test for single leg heel raise | 4 weeks
Change in strength from baseline with the Muscle Endurance Test for single leg heel raise | 3 months

SECONDARY OUTCOMES:
Age | baseline
  Demographic information -
Height | baseline
  Demographic information
Weight | baseline
  Demographic information
Gender | baseline
  Demographic information
Duration of Pain | baseline
  Demographic information

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cleland, DPT, PhD, Study Chair — Nova Southeastern University
Locations (1):
- Breakthrough Physical Therapy, Fayetteville, North Carolina, United States

REFERENCES:
- [Background] Carcia CR, Martin RL, Houck J, Wukich DK; Orthopaedic Section of the American Physical Therapy Association. Achilles pain, stiffness, and muscle power deficits: achilles tendinitis. J Orthop Sports Phys Ther. 2010 Sep;40(9):A1-26. doi: 10.2519/jospt.2010.0305. No abstract available. PMID 20805627
- [Background] Ga H, Choi JH, Park CH, Yoon HJ. Dry needling of trigger points with and without paraspinal needling in myofascial pain syndromes in elderly patients. J Altern Complement Med. 2007 Jul-Aug;13(6):617-24. doi: 10.1089/acm.2006.6371. PMID 17718644
- [Background] Fernandez-Carnero J, La Touche R, Ortega-Santiago R, Galan-del-Rio F, Pesquera J, Ge HY, Fernandez-de-Las-Penas C. Short-term effects of dry needling of active myofascial trigger points in the masseter muscle in patients with temporomandibular disorders. J Orofac Pain. 2010 Winter;24(1):106-12. PMID 20213036
- [Background] Gonzalez-Iglesias J, Cleland JA, del Rosario Gutierrez-Vega M, Fernandez-de-las-Penas C. Multimodal management of lateral epicondylalgia in rock climbers: a prospective case series. J Manipulative Physiol Ther. 2011 Nov;34(9):635-42. doi: 10.1016/j.jmpt.2011.09.003. Epub 2011 Oct 21. PMID 22018577
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Cotchett MP, Munteanu SE, Landorf KB. Effectiveness of trigger point dry needling for plantar heel pain: a randomized controlled trial. Phys Ther. 2014 Aug;94(8):1083-94. doi: 10.2522/ptj.20130255. Epub 2014 Apr 3. PMID 24700136
- [Background] Llamas-Ramos R, Pecos-Martin D, Gallego-Izquierdo T, Llamas-Ramos I, Plaza-Manzano G, Ortega-Santiago R, Cleland J, Fernandez-de-Las-Penas C. Comparison of the short-term outcomes between trigger point dry needling and trigger point manual therapy for the management of chronic mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Nov;44(11):852-61. doi: 10.2519/jospt.2014.5229. Epub 2014 Sep 30. PMID 25269764
- [Background] Osborne NJ, Gatt IT. Management of shoulder injuries using dry needling in elite volleyball players. Acupunct Med. 2010 Mar;28(1):42-5. doi: 10.1136/aim.2009.001560. PMID 20351377
- [Background] Jayaseelan DJ, Moats N, Ricardo CR. Rehabilitation of proximal hamstring tendinopathy utilizing eccentric training, lumbopelvic stabilization, and trigger point dry needling: 2 case reports. J Orthop Sports Phys Ther. 2014 Mar;44(3):198-205. doi: 10.2519/jospt.2014.4905. Epub 2013 Nov 21. PMID 24261928
- [Derived] Koszalinski A, Flynn T, Hellman M, Cleland JA. Trigger point dry needling, manual therapy and exercise versus manual therapy and exercise for the management of Achilles tendinopathy: a feasibility study. J Man Manip Ther. 2020 Sep;28(4):212-221. doi: 10.1080/10669817.2020.1719299. Epub 2020 Feb 12. PMID 32048918